CLINICAL TRIAL: NCT06862518
Title: Ultrasound Guided Serratus Anterior Plane Block Versus Thoracic Erector Spinae Plane Block for Post Operative Analgesia in Pediatrics Undergoing Thoracotomy: A Randomized Controlled Stud
Brief Title: Ultrasound Guided Serratus Anterior Plane Block Versus Thoracic Erector Spinae Plane Block for Post Operative Analgesia in Pediatrics Undergoing Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sarah Elsayed Mohamed Mohamed Hassan, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS209/6/23
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Ultrasound; Serratus Anterior Plane Block; Thoracic Erector Spinae Plane Block; Post Operative Analgesia; Pediatrics; Thoracotomy
MeSH Terms: interventions — Control Groups; Anesthesia, General; Saposins; Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Patients will receive general anesthesia alone
  Interventions: Drug: Control group
- Serratus Anterior Plane Block (SAPB) group (Experimental): Patients will receive general anesthesia (GA) with ultrasound guided serratus anterior plane block 0.5 ml/kg 0.25% bupivacaine.
  Interventions: Drug: Serratus Anterior Plane Block (SAPB) group
- Erector Spinae Plane Block (ESPB) group (Experimental): Patients will receive general anesthesia (GA) with ultrasound guided erector spinae plane block 0.5 ml/kg 0.25% bupivacaine.
  Interventions: Drug: Erector Spinae Plane Block (ESPB) group

INTERVENTIONS:
Drug: Control group — Patients will receive general anesthesia alone
  Other Names: General anesthesia
  Arms: Control group
Drug: Serratus Anterior Plane Block (SAPB) group — Patients will receive general anesthesia (GA) with ultrasound guided serratus anterior plane block 0.5 ml/kg 0.25% bupivacaine.
  Other Names: General anesthesia (GA) with bupivacaine
  Arms: Serratus Anterior Plane Block (SAPB) group
Drug: Erector Spinae Plane Block (ESPB) group — Patients will receive general anesthesia (GA) with ultrasound guided erector spinae plane block 0.5 ml/kg 0.25% bupivacaine
  Other Names: General anesthesia (GA) with bupivacaine
  Arms: Erector Spinae Plane Block (ESPB) group

SUMMARY:
This study is designed to compare the post operative analgesic effect of serratus anterior plane block versus thoracic erector spinae plane block in pediatrics undergoing thoracotomy

DETAILED DESCRIPTION:
The incidence of diseases that requires thoracotomy is low in the pediatric age group. Thoracotomy is a severe burden on children and is widely known to cause severe acute pain. This pain can be very distressing for both children and their parents. If not treated properly, it may acutely cause retention of secretion, atelectasis, ventilation-perfusion disorder and hypoxemia, together with a change in lung mechanics.

The serratus anterior plane block (SAPB) has also recently become more popular options for post-thoracotomy analgesia. SAPB involves local anesthetic injection in a plane superficial or deep to the serratus anterior muscle; in both these locations, it blocks the lateral cutaneous branches of intercostal nerves.

The erector spinae plane block (ESPB) is an ultrasound-guided deep plane interfascial block defined by Forero in 2016. It has been shown to provide thoracic and abdominal analgesia. When injected at the T5 transverse process level, the local anesthetic spreads anteriorly through the thoracolumbar fascia and reaches the ventral and dorsal rami of the spinal nerves and posteriorly to the gray and white rami communicantes of the sympathetic chain, providing a C7 to T8 sensitive block. Although it was first described as a chronic pain block, there are increasingly reports about its use in postoperative acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 2 and 7 years.
* Patient posted for the right or left thoracotomy under general anesthesia.

Exclusion Criteria:

* Parents who refuse regional anesthesia.
* Children who had any coagulation abnormality.
* Deformity of the thoracolumbar spine.
* Infection at the site of injection.
* History of allergy to the local anesthetics.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Total rescue analgesia consumption | 24 hours postoperatively
  Rescue analgesia is planned based on the patients' face, leg, activity, cry, consolability score (FLACC) scores. Morphine 0.05 mg/kg IV was given as rescue analgesia in the case of FLACC scores above 3.The analgesic requirements in the first 24 h postoperatively were recorded.

SECONDARY OUTCOMES:
Time to 1st rescue analgesic requirement | 24 hours postoperatively
  Time to 1st request for the rescue of analgesia (time from the end of surgery till first dose of morphine administrated) was recorded.
Degree of pain | 24 hours postoperatively
  Pain was assessed after surgery over 24 hours using face, leg, activity, cry, consolability score (FLACC) score at following times: 0 (baseline), 1, 3, 6, 8, 12, and 24 h postoperative. FLACC score is used for pain assessment. (Face, legs, activity, cry and Consolability) is a measurement used to assess pain in children between age of 2 to 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0 to 10 with 0 representing no pain, 10 representing the maximum and we start to give rescue analgesia at score 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.